CLINICAL TRIAL: NCT06092788
Title: Phase 1, Randomised, Open-label, 3-way Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics (With Food Effect), and Relative Bioavailability of NTP42:KVA4 Given as a Capsule, Compared With a Liquid, in Healthy Volunteers
Brief Title: Safety, Pharmacokinetics (PK) and Relative Bioavailability of NTP42:KVA4 as a Solid Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ATXA Therapeutics Limited (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATXA-CT002
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTP42:KVA4 Capsule (Experimental)
  Interventions: Drug: NTP42:KVA4 Capsule
- NTP42:KVA4 Oral Suspension (Active Comparator)
  Interventions: Drug: NTP42:KVA4 Liquid

INTERVENTIONS:
Drug: NTP42:KVA4 Capsule — Single doses of NTP42:KVA4 administered to healthy volunteers as a capsule
  Arms: NTP42:KVA4 Capsule
Drug: NTP42:KVA4 Liquid — Single doses of NTP42:KVA4 administered to healthy volunteers as a liquid
  Arms: NTP42:KVA4 Oral Suspension

SUMMARY:
This Phase 1 clinical trial will assess the safety, tolerability and pharmacokinetics (PK) of a solid capsule form of NTP42:KVA4 in male and female healthy volunteers. In a randomised, 3-way cross-over study, the Trial will involve 3 dose sessions where all volunteers will receive 3 single doses of NTP42:KVA4. In two of the dose sessions, volunteers will be fasted where, in one, they will be given the NTP42:KVA4 capsule and, in another, they will be given NTP42:KVA4 in oral liquid form. To test the effect of food on drug absorption (PK), the volunteers will also be given the NTP42:KVA4 capsule after eating a full breakfast.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) in the range 18.0-30.0
* Ability & willingness to provide written consent

Exclusion Criteria:

* Clinically relevant abnormal medical history, physical findings, laboratory values at pre-trial screening.
* History of bleeding disorders, coagulation variables or abnormal blood cell count.
* History of chronic illness.
* Impaired endocrine, thyroid, hepatic, renal or respiratory function, diabetes mellitus, coronary heart disease or history of any psychotic mental illness.
* History of adverse reaction or allergy to any drug.
* Use of aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs), or any other medicine that affects platelet function or coagulation, or any prescription medicine, during the 28 days before the first dose of trial medication.
* History of drug or alcohol abuse
* Smoker or use of nicotine-containing products
* Blood pressure or heart rate at screening outside normal ranges.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of NTP42:KVA4 when given as a capsule in healthy volunteers | Up to 48-hour post-dose
  Adverse events (AEs)
Evaluation of the pharmacokinetics of NTP42:KVA4 when given as a capsule in healthy volunteers | Predose, 0.75-, 2-, 4, 6-, 8-, 12-, 24- & 48-hours post-dosing
  Pharmacokinetic parameter: Area under the curve (AUC)
Evaluation of the effect of food on the pharmacokinetics of NTP42:KVA4 when given as a capsule in healthy volunteers | Predose, 0.75-, 2-, 4, 6-, 8-, 12-, 24- & 48-hours post-dosing
  Pharmacokinetic parameter: Area under the curve (AUC)

SECONDARY OUTCOMES:
Evaluation of the pharmacodynamics effects of NTP42:KVA4 when given as a capsule in healthy volunteers | Predose, 2-, 6-, 24- & 48-hours post-dosing
  TXA2-induced platelet aggregometry

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Yamamoto, MD, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom